CLINICAL TRIAL: NCT07271745
Title: Multicenter Study on Early Arterial Changes in Prediabetic Patients Evaluated by Ultra-High-Frequency Ultrasound（MAP-UHF Study）
Brief Title: Multicenter Study on Early Arterial Changes in Prediabetic Patients Evaluated by Ultra-High-Frequency Ultrasound
Acronym: MAP-UHF
Status: Not yet recruiting | Type: Observational
Sponsor: Chunyan Ma (Other)
Collaborators: Henan Provincial People's Hospital (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor-Investigator, Chunyan Ma, Chief of Cardiovascular Ultrasound, First Hospital of China Medical University
Organization: First Hospital of China Medical University (Other)
Other Study IDs: MAP-UHF-01
Record Dates: First submitted 2025-08-20; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Prediabetes
Keywords: Ultra-High-Frequency Ultrasound; Prediabetic; Arterial Changes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy control group: According to the criteria for establishing normal values, a total of 1,440 healthy Chinese adults were enrolled, stratified by gender and age, with 720 males and 720 females.
- Prediabetic Patients group: Patients meeting the 2019 WHO diagnostic criteria for prediabetes: impaired fasting glucose (venous plasma glucose ≥6.1 mmol/L, <7.0 mmol/L, and <7.8 mmol/L after glucose loading) and/or impaired glucose tolerance (venous plasma glucose <7.0 mmol/L, and ≥7.8 mmol/L, <11.1 mmol/L after glucose loading).
  A total of 300 prediabetic patients were included.

SUMMARY:
Ultra-high frequency ultrasound technology (20-100 MHz) can clearly distinguish the arterial intima and media layers, and can simultaneously meet the needs of examining the carotid artery and peripheral arteries, enabling earlier and more accurate detection of vascular damage in pre-diabetic individuals. Therefore, this study aims to establish the normal values of arterial intima and media thickness measured by ultra-high frequency ultrasound in healthy Chinese adults, providing quantitative reference for the early diagnosis, severity assessment, and efficacy observation of arterial diseases. Meanwhile, by applying ultra-high frequency ultrasound, this study intends to clarify the changes in arterial intima and media thickness in pre-diabetic populations and explore the influencing factors, so as to provide reference for the early prevention, diagnosis, and treatment of pre-diabetes and cardiovascular complications.

DETAILED DESCRIPTION:
The arterial wall consists of the intima, media, and adventitia from inside to outside. Among them, intima-media thickness (IMT) is an important criterion for reflecting subclinical arteriosclerosis. However, this composite index has certain limitations. The pathological changes of atherosclerosis mainly occur in the intima, while hypertension, diabetes, etc., mainly affect the media. Therefore, measuring the thickness of the arterial intima and media separately can reflect the degree of vascular lesions in different diseases earlier and more accurately than IMT, which is of great clinical significance. However, there are currently no normal reference values for the thickness of the arterial intima and media.

Diabetes is one of the fastest-growing global public health events in the 21st century, with its prevalence and mortality rate ranking among the top of various diseases. Diabetes is also one of the diseases with the most complications, among which cardiovascular complications cause the greatest harm to patients and have become the leading cause of death in such patients. The vast majority of patients go through a pre-diabetic stage before developing clinically diagnosed diabetes. Epidemiological survey results show that the number of patients in the pre-diabetic stage is much larger than that of diabetic patients. In addition, before diabetes is diagnosed, hyperglycemia may have already caused vascular damage, first leading to thickening and calcification of the arterial media. Studies have shown that the prevalence of vascular calcification in pre-diabetic patients is much higher than that in non-diabetic patients. Early detection of medial vascular calcification is of great clinical value for evaluating vascular changes in pre-diabetes and thus enabling early prevention. However, there is a lack of relevant studies confirming the vascular lesions in pre-diabetes.

In the past, the ultrasound probes used for clinical examination of the carotid artery and peripheral arteries were mainly 5-10 MHz, with a resolution of 200-400 μm, which cannot clearly display the fine structure of the arterial wall, making it difficult to measure the intima or media alone. With the development of modern medical technology, the emergence of ultra-high frequency ultrasound (20-100 MHz) can clearly distinguish the arterial intima and media, and can simultaneously meet the needs of examining the carotid artery and peripheral arteries. It is expected to reflect vascular lesions caused by different diseases more sensitively and accurately, providing a new and beneficial tool for clinical observation of arterial structure.

In recent years, the ultra-high frequency ultrasound technology (20-100 MHz) has emerged, which can clearly distinguish the arterial intima and media, and can simultaneously meet the needs of examining the carotid artery and peripheral arteries, enabling earlier and more accurate detection of vascular damage in pre-diabetes. Therefore, our center has initiated this multi-center clinical research project, joining hands with multiple ultrasound centers across the country, aiming to establish the normal values of arterial intima and media thickness measured by ultra-high frequency ultrasound in healthy Chinese adults, providing quantitative reference for the early diagnosis, degree assessment, and efficacy observation of arterial diseases. At the same time, it aims to use ultra-high frequency ultrasound to clarify the changes in arterial intima and media thickness in pre-diabetic populations, explore the influencing factors, and provide reference for the early prevention, diagnosis, and treatment of pre-diabetes and cardiovascular complications.

ELIGIBILITY:
Prediabetic Patients

Inclusion Criteria:

* Impaired fasting glucose (venous plasma glucose ≥6.1 mmol/L, <7.0 mmol/L, and <7.8 mmol/L 2 hours after glucose loading); and/or Impaired glucose tolerance (venous plasma glucose <7.0 mmol/L, and ≥7.8 mmol/L, <11.1 mmol/L 2 hours after glucose loading).
* Age ≥ 18 years old;
* Normal blood pressure (139-90/89-60 mmHg);
* Body mass index (BMI) < 30 kg/m²;
* Normal results in routine blood tests, fasting blood glucose, lipid profile, liver and kidney function tests, and electrocardiogram (ECG);
* No history of cardiovascular diseases, diabetes, rheumatic connective tissue diseases, or severe liver/kidney dysfunction;
* No history of acrocyanosis, no discomfort under cold stimulation, and no previous Raynaud's phenomenon in any part of the body;
* No history of taking medications that affect the cardiovascular system.

Exclusion Criteria :

* Patients with hypertension, diabetes mellitus, hyperthyroidism, arrhythmia, etc.
* Patients with connective tissue diseases such as systemic lupus erythematosus, polymyositis, rheumatoid arthritis, etc.
* History of blood diseases, severe infections, or other systemic diseases.
* Administration of vasoactive drugs within the past month.
* Peripheral vascular diseases with arterial occlusion that prevents detection of blood flow signals.
* Inability to cooperate with the examination.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 300 prediabetic patients were selected from the physical examination center and outpatient department, and 1,440 healthy subjects were enrolled.
Sampling Method: Probability Sample
Enrollment: 1740 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the thickness of the arterial intima (mm), media (mm), and intima-media (mm) respectively | 1 day
  Measuring the thickness of the arterial intima and media separately can more early and accurately reflect the degree of vascular lesions in different diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ma, Ph.D., Principal Investigator — First Hospital of China Medical University
Locations (30):
- China (30):
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi University of Chinese Medicine, Nanning, Guangxi
  - The First Affiliated Hospital of Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Second Hospital of Heilongjiang Province, Harbin, Heilongjiang
  - Jiamusi Central Hospital, Heilongjiang Province, Jiamusi, Heilongjiang
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jinlin
  - The First Hospital of Jilin University, Changchun, Jinlin
  - Anshan Central Hospital, Anshan, Liaoning
  - Chaoyang Central Hospital, Chaoyang, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - Tongliao People's Hospital of Inner Mongolia Autonomous Region, Tongliao, Neimenggu
  - Qilu Hospital (Qingdao Branch) of Shandong University, Qingdao, Shandong
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Third People's Hospital of Yunnan Province, Kunming, Yunnan
  - The Second People's Hospital of Qujing City, Qujing, Yunnan
  - Li Huili Hospital of Ningbo Medical Center, Zhejiang Province, Ningbo, Zhejing
  - Beijing Hospital, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Jiading District Central Hospital of Shanghai Municipality, Shanghai
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Yueyang Hospital of Integrated Traditional Chinese and Western Medicine Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai
  - The Third Central Hospital of Tianjin, Tianjin

IPD SHARING:
Plan to Share IPD: No